CLINICAL TRIAL: NCT06235645
Title: dEtection of rheumAtoid aRthritis - Interstitial Lung dIseasE by Thoracic ultRasound
Acronym: EARLIER
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: DR230226 - EARLIER
Record Dates: First submitted 2024-01-23; First posted 2024-02-01 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Rheumatoid Arthritis; Interstitial Lung Disease; Thoracic Ultrasound; Lung Ultrasound
Keywords: Lung ultrasound; Rheumatoid Arthritis; Interstitial Lung Disease
MeSH Terms: conditions — Arthritis, Rheumatoid; Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Lung ultrasound (LUS) — If included, an LUS will be performed by an experienced operator, blinded to the results of the chest CT and PFT.
  A linear probe (4 to 12 MHz) will be used. The patient will be installed́ in a semi-seated position with the homolateral arm above the head for the anterior and axillary evaluation then, depending on his comfort, in a seated position or in right then left lateral decubitus, arms alongside the body, for the posterior evaluation. It will be practiced by experienced operators (pneumologist) and according to a validated protocol allowing the exploration of 14 intercostal spaces. LUT will be timed, recorded and anonymized.
  The operator will note the 3 ultrasound signs (total number of B lines, pleural line thickening and percentage of pleural line irregularity), their location and severity.
  The radiologist, on his part, will evaluate the patient's chest CT (gold standard), blinded to the results of the LUS, to make or not the diagnosis of RA-ILD.

SUMMARY:
Rheumatoid arthritis is an autoimmune disease that can affect various organs, including the lungs, and lead to rheumatoid arthritis-interstitial lung disease (RA-ILD).

RA-ILD is responsible for increased mortality in rheumatoid arthristis (RA) patients.

The prevalence of RA-ILD varies according to the screening tool used.

The current gold standard is chest CT, but this is an expensive, time-consuming and irradiating examination, and recommendations on when and how often it should be performed are not clearly established.

Lung ultrasound (LUS) is an emerging tool for the detection of lung parenchymal damage, particularly in systemic scleroderma and idiopathic pulmonary fibrosis (IPF).

LUS is a non-irradiating, non-expensive examination that can be performed rapidly.

The aim of our study is to evaluate LUS as a screening tool for RA-ILD, in patients with risk factors for developing RA-ILD.

DETAILED DESCRIPTION:
Patients with RA and who have risk factors for RA-ILD are regularly reassessed in a rheumatology day hospital.

As part of their routine follow-up, and given the absence of recommendations on screening for RA-ILD in this population, chest CT and PFT (pulmonary function tests) are regularly performed at the request of the rheumatologist.

Therefore, all patients meeting the inclusion criteria and having undergone chest CT and PFT in the 6 months preceding or following their rheumatology reassessment will be offered participation in the study.

Participation in the study does not alter the patient's usual follow-up.

Objective of the study: evaluate the sensitivity and specificity of thoracic ultrasound compare to the chest CT in patients with risk factors of developing RA-ILD.

Design: This is a non-interventional, prospective, single-center, multidisciplinary study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (age > 18 years) followed at CHU of Tours
* Diagnosis of rheumatoid arthritis validated according to ACR 2010 criteria, EULAR classification, regardless of time since diagnosis
* Patient who has had or will have a thoracic CT scan and PFT performed as part of routine care in the 6 months preceding or following inclusion
* Patient with at least two risk factors for developing RA-ILD among :

  * Male sex or
  * Active or former smoker assessed at 20 pack-year or
  * Age > 60 years or
  * Levels of RF≥3N (rheumatoid factor) and/or anti-CCP≥3N (antibodies against cyclic citrullinated peptides) at diagnosis or at any time during the course of the disease or
  * High RA activity score (DAS28>3.2)

Exclusion Criteria:

* Diagnosis of congenital lung disease
* Diagnosis of another autoimmune pathology associated with RA (overlap syndrome) linked to the development of ILD (interstitial lung disease) (systemic sclerosis, myositis, dermatomyositis, mixed connectivitis, systemic lupus erythematosus or other ANCA vasculitis, with the exception of secondary Gougerot-Sjögren's syndromes).
* Current or operated lung cancer
* Thoracic irradiation
* Thoracic transplant patients
* Previous invasive thoracic procedures
* Pathologies responsible for pleural thickening (silicosis, asbestosis, known pleural plaque, pleural sequelae of tuberculosis)
* Pregnant or breast-feeding women
* Patient under legal protection (guardianship, curatorship or safeguard of justice)
* Patient who has objected to data processing
* Parenchymal infection current or less than one month old prior to LUS examination
* Liquid or gaseous pleural effusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients followed at CHU de Tours with a diagnosis of rheumatoid arthritis and with at least two risk factors for developing PR-PID
Sampling Method: Non-Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Determination sensitivity and specificity of thoracic ultrasound | 2 years
  The primary outcome is to determine the sensitivity and specificity of thoracic ultrasound defined as pathological by a total number of B lines ≥ 9 and/or pleural line thickening ≥ 3mm and/or a percentage of pleural line irregularity ≥ 24%.

SECONDARY OUTCOMES:
Percentage of each of the 3 ultrasound signs among pathological ultrasounds. | 2 years
  The secondary outcome is the percentage of each of the 3 ultrasound signs among pathological ultrasounds.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie LEGUE, Principal Investigator — University Hospital, Tours
Locations (1):
- university hospital Tours, Tours, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Gabbay E, Tarala R, Will R, Carroll G, Adler B, Cameron D, Lake FR. Interstitial lung disease in recent onset rheumatoid arthritis. Am J Respir Crit Care Med. 1997 Aug;156(2 Pt 1):528-35. doi: 10.1164/ajrccm.156.2.9609016. PMID 9279235
- [Result] Olson AL, Swigris JJ, Sprunger DB, Fischer A, Fernandez-Perez ER, Solomon J, Murphy J, Cohen M, Raghu G, Brown KK. Rheumatoid arthritis-interstitial lung disease-associated mortality. Am J Respir Crit Care Med. 2011 Feb 1;183(3):372-8. doi: 10.1164/rccm.201004-0622OC. Epub 2010 Sep 17. PMID 20851924
- [Result] Hyldgaard C, Hilberg O, Pedersen AB, Ulrichsen SP, Lokke A, Bendstrup E, Ellingsen T. A population-based cohort study of rheumatoid arthritis-associated interstitial lung disease: comorbidity and mortality. Ann Rheum Dis. 2017 Oct;76(10):1700-1706. doi: 10.1136/annrheumdis-2017-211138. Epub 2017 Jun 13. PMID 28611082
- [Result] Brown KK. Rheumatoid lung disease. Proc Am Thorac Soc. 2007 Aug 15;4(5):443-8. doi: 10.1513/pats.200703-045MS. PMID 17684286
- [Result] Bongartz T, Nannini C, Medina-Velasquez YF, Achenbach SJ, Crowson CS, Ryu JH, Vassallo R, Gabriel SE, Matteson EL. Incidence and mortality of interstitial lung disease in rheumatoid arthritis: a population-based study. Arthritis Rheum. 2010 Jun;62(6):1583-91. doi: 10.1002/art.27405. PMID 20155830
- [Result] Chen J, Shi Y, Wang X, Huang H, Ascherman D. Asymptomatic preclinical rheumatoid arthritis-associated interstitial lung disease. Clin Dev Immunol. 2013;2013:406927. doi: 10.1155/2013/406927. Epub 2013 Jul 31. PMID 23983768
- [Result] Dawson JK, Fewins HE, Desmond J, Lynch MP, Graham DR. Fibrosing alveolitis in patients with rheumatoid arthritis as assessed by high resolution computed tomography, chest radiography, and pulmonary function tests. Thorax. 2001 Aug;56(8):622-7. doi: 10.1136/thorax.56.8.622. PMID 11462065
- [Result] Matson S, Lee J, Eickelberg O. Two sides of the same coin? A review of the similarities and differences between idiopathic pulmonary fibrosis and rheumatoid arthritis-associated interstitial lung disease. Eur Respir J. 2021 May 13;57(5):2002533. doi: 10.1183/13993003.02533-2020. Print 2021 May. PMID 33303554
- [Result] Kawano-Dourado L, Doyle TJ, Bonfiglioli K, Sawamura MVY, Nakagawa RH, Arimura FE, Lee HJ, Rangel DAS, Bueno C, Carvalho CRR, Sabbag ML, Molina C, Rosas IO, Kairalla RA. Baseline Characteristics and Progression of a Spectrum of Interstitial Lung Abnormalities and Disease in Rheumatoid Arthritis. Chest. 2020 Oct;158(4):1546-1554. doi: 10.1016/j.chest.2020.04.061. Epub 2020 May 16. PMID 32428513
- [Result] Zamora-Legoff JA, Krause ML, Crowson CS, Ryu JH, Matteson EL. Progressive Decline of Lung Function in Rheumatoid Arthritis-Associated Interstitial Lung Disease. Arthritis Rheumatol. 2017 Mar;69(3):542-549. doi: 10.1002/art.39971. PMID 27788297
- [Result] Mohammadi A, Oshnoei S, Ghasemi-rad M. Comparison of a new, modified lung ultrasonography technique with high-resolution CT in the diagnosis of the alveolo-interstitial syndrome of systemic scleroderma. Med Ultrason. 2014 Mar;16(1):27-31. doi: 10.11152/mu.2014.2066.161.am1so2. PMID 24567921
- [Result] Manolescu D, Oancea C, Timar B, Traila D, Malita D, Birsasteanu F, Tudorache V. Ultrasound mapping of lung changes in idiopathic pulmonary fibrosis. Clin Respir J. 2020 Jan;14(1):54-63. doi: 10.1111/crj.13101. Epub 2019 Nov 14. PMID 31675455
- [Result] Pinal-Fernandez I, Pallisa-Nunez E, Selva-O'Callaghan A, Castella-Fierro E, Simeon-Aznar CP, Fonollosa-Pla V, Vilardell-Tarres M. Pleural irregularity, a new ultrasound sign for the study of interstitial lung disease in systemic sclerosis and antisynthetase syndrome. Clin Exp Rheumatol. 2015 Jul-Aug;33(4 Suppl 91):S136-41. Epub 2015 Aug 27. PMID 26315813
- [Result] Gutierrez M, Tardella M, Rodriguez L, Mendoza J, Clavijo-Cornejo D, Garcia A, Bertolazzi C. Ultrasound as a potential tool for the assessment of interstitial lung disease in rheumatic patients. Where are we now? Radiol Med. 2019 Oct;124(10):989-999. doi: 10.1007/s11547-019-01053-5. Epub 2019 Jul 2. PMID 31267321
- [Result] Cogliati C, Antivalle M, Torzillo D, Birocchi S, Norsa A, Bianco R, Costantino G, Ditto MC, Battellino M, Sarzi Puttini PC, Montano N. Standard and pocket-size lung ultrasound devices can detect interstitial lung disease in rheumatoid arthritis patients. Rheumatology (Oxford). 2014 Aug;53(8):1497-503. doi: 10.1093/rheumatology/keu033. Epub 2014 Mar 31. PMID 24692573